CLINICAL TRIAL: NCT05613569
Title: A Long-term, 3-Year, Follow-up Study for Patients Completing the KS-GIG-001-01 Study
Status: Active, not recruiting | Type: Observational
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Other Study IDs: KLS-2031LSRL001
Record Dates: First submitted 2022-10-07; First posted 2022-11-14 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Lumbosacral Radiculopathy
Keywords: Lumbosacral Radiculopathy; LSR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: KLS-2031 — KLS-2031 administered by transforaminal epidural injection

SUMMARY:
This is a long-term, 3-year, follow-up study for patients completing the KS-GIG-001-01 Study

DETAILED DESCRIPTION:
This is a long-term, 3-year, follow-up study for patients completing the KS-GIG-001-01 Study (A Phase 1/2a, First-in-Human, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Therapeutic Activity of Single Ascending Doses of KLS-2031 Administered by Transforaminal Epidural Injection in Patients with Neuropathic Pain from Lumbosacral Radiculopathy). Following the end of the Open-label Safety Extension Period of the KS-GIG-001-01 Study (Visit 14), patients will enter the Long-term Follow-up Period. These patients will continue to be monitored for AEs (including AEs of special interest) and serious AEs (SAEs) via phone call every 6 months and outpatient visits every 52 weeks (annually), over 3 years.

ELIGIBILITY:
Inclusion Criteria :

To be considered eligible to participate in this study, a patient must meet the inclusion criteria listed below:

1. Patients that have completed the KS-GIG-001-01 Study and were in the Active Treatment group
2. Patients having signed the consent forms for both the KS-GIG-001-01 Study and this Long Term, 3-Year Follow-up Study

Exclusion Criteria :

To be eligible for entry into the study, the patient must not meet any of the exclusion criteria listed below:

1. Enrollment in another AAV or other gene therapy trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This long-term follow-up study will include up to 12 patients with neuropathic pain from LSR that have completed the KS-GIG-001-01 Study and were randomized to receive KLS-2031.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of KLS-2031 as assessed by frequency and nature of AEs, laboratory test results, vital sign measurements, physical and complete neurological examinations, and 12 lead ECGs through 156 weeks. | Baseline through the end of study (approximately 3 years)
  Long-term safety of KLS-2031 as assessed by frequency and nature of AEs, laboratory test results, vital sign measurements, physical and complete neurological examinations, and 12 lead ECGs through 156 weeks.

SECONDARY OUTCOMES:
Change from baseline to each visit in Pain Intensity Numerical Rating Scale (PI-NRS) score = Result at week n - baseline, (n=52, 104, 156) | Week 52, Week 104, Week 156
  The PI-NRS is measured on an 11-point numerical scale ranging from 0 (no pain) to 10 (worst possible pain) that the patient selects to best describe the intensity of pain that they have experienced in the last 24 hours.
Change from baseline to each visit in Daily Sleep Interference Scale (DSIS) score = Result at week n - baseline, (n=52, 104, 156) | Week 52, Week 104, Week 156
  The DSIS has an 11-point numerical scale that asks the patient to assess how pain has interfered with their sleep during the past 24 hours. Response options range from 0 (does not interfere with sleep) to 10 (completely interferes with sleep).
Change from baseline to each visit in Galer Neuropathic Pain Scale (Galer NPS) score = Result at week n - baseline, (n=52, 104, 156) | Week 52, Week 104, Week 156
  The Galer NPS is a relatively simple, self-administered, 10-item questionnaire for evaluating pain, which assesses distinct pain qualities associated with neuropathic pain.
Change from baseline to each visit in modified Roland-Morris Disability Questionnaire (RMDQ) score = Result at week n - baseline, (n=52, 104, 156) | Week 52, Week 104, Week 156
  The modified RMDQ is a self-administered, 24-question physical disability measurement tool that evaluates both back and leg pain. Each of the 24 questions is asked 2 times, once with regard to back pain and once with regard to leg pain, for a total of 48 items. Each question requires a "yes" or "no" answer; 1 point is scored for each positive response. The total scores are determined on a scale of 0 to 24 for back pain and on a scale of 0 to 24 for leg pain, with 0 representing "no disability" and 24 representing "extreme disability."

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- Kolon Investigative Site : CenExel JBR, Salt Lake City, Utah, United States